CLINICAL TRIAL: NCT02507687
Title: A Comparison of Bimatoprost SR to Selective Laser Trabeculoplasty in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Comparison of Bimatoprost Sustained Release (SR) to Selective Laser Trabeculoplasty (SLT) in Adults With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192024-093; 2015-002131-18 (EudraCT Number)
Expanded Access: NCT05338606 (No longer available)
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Results first posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-04

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Stage 1: SLT (Primary Eye) / Bimatoprost SR 15 µg (Contralateral Eye) (Experimental): Participants enrolled prior to implementation of Protocol Amendment 3 receive the following treatment in each eye:
  Assigned Primary Eye: Selective laser trabeculoplasty (SLT) administered on Day 1 followed by up to three sham bimatoprost SR administrations.
  Contralateral Eye: Sham SLT administered on Day 1 followed by up to three bimatoprost SR 15 µg administrations.
  Bimatoprost SR/sham bimatoprost SR is administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2) and Week 32 (Cycle 3; participants who reach Week 32 prior to implementation of Protocol Amendment 3 only).
  Interventions: Drug: Bimatoprost SR; Drug: Sham Bimatoprost SR; Procedure: Selective Laser Trabeculoplasty; Procedure: Sham Selective Laser Trabeculoplasty
- Stage 1: Bimatoprost SR 15 µg (Primary Eye) / SLT (Contralateral Eye) (Experimental): Participants enrolled prior to implementation of Protocol Amendment 3 receive the following treatment in each eye:
  Assigned Primary Eye: Sham SLT administered on Day 1 followed by up to three bimatoprost SR 15 µg administrations.
  Contralateral Eye: SLT administered on Day 1 followed by up to three sham bimatoprost SR administrations.
  Bimatoprost SR/sham bimatoprost SR is administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2) and Week 32 (Cycle 3; participants who reach Week 32 prior to implementation of Protocol Amendment 3 only).
  Interventions: Drug: Bimatoprost SR; Drug: Sham Bimatoprost SR; Procedure: Selective Laser Trabeculoplasty; Procedure: Sham Selective Laser Trabeculoplasty
- Stage 2: SLT (Primary Eye) / Bimatoprost SR 10 µg (Contralateral Eye) (Experimental): Participants enrolled after implementation of Protocol Amendment 3 receive the following treatment in each eye:
  Assigned Primary Eye: SLT administered on Day 1 followed by up to two sham bimatoprost SR administrations.
  Contralateral Eye: Sham SLT administered on Day 1 followed by up to two bimatoprost SR 10 µg administrations.
  Bimatoprost SR/sham bimatoprost SR is administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2). After implementation of Protocol Amendment 6, Cycle 2 retreatment could occur after Week 16 and prior to Month 12 based on when retreatment criteria are met.
  Interventions: Drug: Bimatoprost SR; Drug: Sham Bimatoprost SR; Procedure: Selective Laser Trabeculoplasty; Procedure: Sham Selective Laser Trabeculoplasty
- Stage 2: Bimatoprost SR 10 µg (Primary Eye) / SLT (Contralateral Eye) (Experimental): Participants enrolled after implementation of Protocol Amendment 3 receive the following treatment in each eye:
  Assigned Primary Eye: Sham SLT administered on Day 1 followed by up to two bimatoprost SR 10 µg administrations.
  Contralateral Eye: SLT administered on Day 1 followed by up to two sham bimatoprost SR administrations.
  Bimatoprost SR/sham bimatoprost SR is administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2). After implementation of Protocol Amendment 6, Cycle 2 retreatment could occur after Week 16 and prior to Month 12 based on when retreatment criteria were met.
  Interventions: Drug: Bimatoprost SR; Drug: Sham Bimatoprost SR; Procedure: Selective Laser Trabeculoplasty; Procedure: Sham Selective Laser Trabeculoplasty

INTERVENTIONS:
Drug: Bimatoprost SR — Bimatoprost SR is a biodegradable, sustained-release, preservative-free bimatoprost implant, preloaded in an applicator for administration. The Bimatoprost SR implant is injected into the anterior chamber via the corneal limbus using the prefilled applicator.
Drug: Sham Bimatoprost SR — Sham bimatoprost SR performed using the same procedure as for Bimatoprost SR using an needleless applicator that touches the eye at the area of insertion but does not deliver an implant into the anterior chamber.
Procedure: Selective Laser Trabeculoplasty — SLT is a laser procedure that targets the melanin, or pigment, in specific cells of the eye.
  An ophthalmologist performed 360 degrees of SLT using a standardized method.
Procedure: Sham Selective Laser Trabeculoplasty — Sham SLT is performed on the contralateral eye using the same method as for SLT, with the exception that the laser is not switched to the active state.

SUMMARY:
This study will evaluate the intraocular pressure (IOP)-lowering effect and safety of bimatoprost SR compared with selective laser trabeculoplasty in patients with open-angle glaucoma or ocular hypertension who are not adequately managed with topical IOP-lowering medication for reasons other than medication efficacy (e.g., due to intolerance or nonadherence).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either open-angle glaucoma or ocular hypertension in each eye that require IOP lowering treatment.
* In the investigator's opinion, patient's IOP is not adequately managed with topical medication for reasons other than medication efficacy (eg, due to intolerance or nonadherence).
* In the investigator's opinion, both eyes can be treated adequately with topical prostamide, prostaglandin, or prostaglandin analog eye drops as the sole therapy if medication was taken as directed, or with SLT monotherapy.

Exclusion Criteria:

* History of previous laser trabeculoplasty
* History or evidence of complicated cataract surgery: eg, surgery resulting in complicated lens placement (such as anterior chamber intraocular lens implant [IOL], sulcus IOL, aphakia, etc) or intraoperative complications (such as a posterior capsular tear [with or without vitreous loss], substantial iris trauma, etc) or history of phakic IOL insertion for refractive error correction
* Intraocular surgery (including cataract surgery) and/or any ocular laser surgery within the 6 months prior to treatment
* Previous use of commercially available Bimatoprost SR; concurrent enrollment in another Allergan Bimatoprost SR study; or previous enrollment in which an implant was received.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (95):
- United States (51):
  - Trinity Research Group /ID# 234598, Dothan, Alabama
  - Arizona Advanced Eye Research Institute /ID# 234947, Glendale, Arizona
  - Arizona Glaucoma Specialists /ID# 235066, Phoenix, Arizona
  - M&M Eye Institute /ID# 235391, Prescott, Arizona
  - Walman Eye Center /ID# 236054, Sun City, Arizona
  - California Center for Clin Res /ID# 237412, Arcadia, California
  - Orange County Ophthalmology /ID# 235995, Garden Grove, California
  - Speciality Eye Care Medical Group /ID# 236001, Glendale, California
  - Lugene Eye Institute /ID# 237042, Glendale, California
  - Lakeside Vision Center /ID# 234971, Irvine, California
  - California Eye Specialists Medical Group Inc. /ID# 235999, Pasadena, California
  - North Bay Eye Associates Inc. /ID# 235429, Petaluma, California
  - Pacific Eye Associates /ID# 235326, San Francisco, California
  - Wolstan & Goldberg Eye Associates /ID# 235166, Torrance, California
  - Segal Drug Trials Inc. /ID# 235169, Delray Beach, Florida
  - Eye Associates of South West Florida /ID# 235424, Fort Myers, Florida
  - Levenson Eye Associates Inc. /ID# 235021, Jacksonville, Florida
  - University of Florida /ID# 236876, Jacksonville, Florida
  - Ocala Eye PA /ID# 235431, Ocala, Florida
  - Dr. Andrew Gardner Logan, FL /ID# 236946, Tamarac, Florida
  - University of South Florida /ID# 237737, Tampa, Florida
  - Clayton Eye Clinical Research, LLC /ID# 236678, Morrow, Georgia
  - University of Illinois at Chicago Illinois Eye and Ear Infirmary /ID# 234875, Chicago, Illinois
  - Sabates Eye Centers /ID# 234868, Leawood, Kansas
  - Cincinnati Eye Institute- Edgewood /ID# 236714, Edgewood, Kentucky
  - The Eye Care Institute /ID# 236690, Louisville, Kentucky
  - Advanced Glaucoma Specialists /ID# 234799, Reading, Massachusetts
  - Fraser Eye Center /ID# 235791, Fraser, Michigan
  - Midwest Vision Research Foundation at Pepose Vision Institute /ID# 235879, Chesterfield, Missouri
  - Northern New Jersey Eye Institute PA /ID# 234944, South Orange, New Jersey
  - Eye Associates of New Mexico /ID# 235115, Albuquerque, New Mexico
  - Albemarle Clinical Trials LLC /ID# 235144, Elizabeth City, North Carolina
  - Duplicate_Cornerstone Eye Care /ID# 235047, High Point, North Carolina
  - Bagan Strinden Vision /ID# 234898, Fargo, North Dakota
  - Oklahoma Eye Surgeons /ID# 235848, Oklahoma City, Oklahoma
  - Scott and Christie and Associates /ID# 234594, Cranberry Township, Pennsylvania
  - Eye Care Specialists /ID# 235129, Kingston, Pennsylvania
  - Family Eye Group P.C. /ID# 236114, Lancaster, Pennsylvania
  - Wills Eye Hospital /ID# 236487, Philadelphia, Pennsylvania
  - Carolinas Centers for Sight,PC /ID# 237017, Florence, South Carolina
  - Chattanooga Eye Institute /ID# 235250, Chattanooga, Tennessee
  - ATX Clinical Trials Inc. dba Keystone Research /ID# 235869, Austin, Texas
  - Cross Eye Center /ID# 236116, Bellaire, Texas
  - Houston Eye Associates /ID# 237883, Houston, Texas
  - Baylor College of Medicine - Baylor Medical Center /ID# 237148, Houston, Texas
  - San Antonio Eye Center /ID# 235632, San Antonio, Texas
  - Eye associates /ID# 236501, San Antonio, Texas
  - Medical Center Ophthalmology Associates /ID# 235016, San Antonio, Texas
  - Emerson Clinical Research Institute /ID# 235977, Falls Church, Virginia
  - Piedmont Eye Center /ID# 234533, Lynchburg, Virginia
  - West Virginia University Eye Institute /ID# 235174, Morgantown, West Virginia
- Australia (8):
  - Queensland Eye Institute /ID# 236074, South Brisbane, Queensland
  - Eye Surgery Associates /ID# 235872, East Melbourne, Victoria
  - Melbourne Eye Specialists /ID# 234614, Fitzroy, Victoria
  - Waverley Eye Clinic /ID# 234997, Glen Waverley, Victoria
  - The Lions Eye Institute /ID# 236832, Nedlands, Western Australia
  - Essendon Eye Clinic /ID# 235433, Essendon
  - Geelong Eye Clinic /ID# 236118, Geelong
  - Vision Eye Institute /ID# 236003, Melbourne
- Ophthalmology Clinic Bellevue /ID# 234631, Montreal, Quebec, Canada
- Rigshospitalet Glostrup /ID# 237709, Glostrup Municipality, Capital Region, Denmark
- France (7):
  - Chu Angers /Id# 237805, Angers
  - Polyclinique de la Baie /ID# 235842, Avranches
  - CHU Bordeaux - Hopital Pellegrin /ID# 237705, Bordeaux
  - Clinique Honore Cave - Pharmacie /ID# 235925, Montauban
  - CHU de Nice - Hospital Pasteur 2 /ID# 235844, Nice
  - CHU Strasbourg - Hopital Civil /ID# 237837, Strasbourg
  - Chu Toulouse Purpan - Hopital Pierre Paul Riquet /ID# 235841, Toulouse
- Germany (3):
  - Internationale Innovative Ophthalmochirurgie /ID# 235263, Düsseldorf, North Rhine-Westphalia
  - Charite Universitaetsklinikum Berlin - Campus Virchow /ID# 235966, Berlin
  - Universitaetsklinikum Magdeburg /ID# 237284, Magdeburg
- Israel (5):
  - Tel Aviv Sourasky Medical Center /ID# 237211, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 237741, Haifa
  - The Lady Davis Carmel Medical Center /ID# 236757, Haifa
  - Galilee Medical Center /ID# 235742, Nahariya
  - Rabin Medical Center /ID# 237698, Petah Tikva
- New Zealand (3):
  - Auckland Eye Hospital /ID# 235253, Remuera, Auckland
  - Southern Eye Specialists /ID# 236081, Christchurch, Canterbury
  - Capital Eye Specialists /ID# 236111, Wellington
- Philippines (4):
  - Asian Eye Institute /ID# 235092, Makati City
  - Peregrine Eye and Laser Institute /ID# 236220, Makati City
  - American Eye Center /ID# 235320, Makati City
  - Cardinal Santos Medical Center /ID# 235325, San Juan City
- Centrum Diagnostyki i Mikrochirurgii Oka - LENS dr n. med. Slawomir Zalewski /ID# 235929, Olsztyn, Poland
- Russia (2):
  - Clinical ophthalmology hospital n.a. V.P. Vihodtsev. /ID# 236041, Omsk
  - Samara State Medical University /ID# 236997, Samara
- United Kingdom (9):
  - University Hospital of Derby and Burton NHS Foundation Trust /ID# 237129, Derby, Derbyshire
  - Queen Mary's Hospital /ID# 234899, Greater London, Kent
  - Guys and St Thomas NHS Foundation Trust /ID# 236806, London, London, City of
  - Epsom & St Helier University Hospital NHS Trust /ID# 236902, Carshalton, Surrey
  - Cambridge University Hospitals NHS Foundation Trust /ID# 238315, Cambridge
  - NHS Lothian /ID# 237450, Edinburgh
  - Moorfields Eye Hospital NHS Foundation Trust /ID# 237708, London
  - Imperial College Healthcare NHS Trust /ID# 234777, London
  - Manchester University NHS Foundation Trust /ID# 237318, Manchester

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Kolko M, Tatham AJ, Lim KS, Wells AP, Shiu M, Uy HS, Sarkisian SR Jr, Ho Q, Jiao J, Kim K, Goodkin ML, Bejanian M, Robinson MR, Paauw JD; ATHENA STUDY GROUP. Phase 3, Randomized, Comparison Study of Intracameral Bimatoprost Implant 10 microg and Selective Laser Trabeculoplasty. Am J Ophthalmol. 2025 Apr;272:19-37. doi: 10.1016/j.ajo.2024.12.026. Epub 2025 Jan 10. PMID 39800203
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=192024-093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 61 sites in 11 countries (Australia, Canada, Germany, Denmark, France, Great Britain, Israel, New Zealand, Philippines, Poland, and the US).
  The eye with the higher intraocular pressure (IOP) at Baseline was assigned as the primary eye. If Baseline IOP was the same in both eyes, the right eye was the primary eye.
Pre-assignment Details: The primary eye was randomized to receive either bimatoprost sustained release (SR) or selective laser trabeculoplasty (SLT) using a 1:1 ratio. If the primary eye received bimatoprost SR, the contralateral eye received SLT. If the primary eye received SLT, the contralateral eye received bimatoprost SR.
Groups:
- Stage 1: SLT (Primary Eye) / Bimatoprost SR 15 µg (Contralateral Eye): Participants enrolled prior to implementation of Protocol Amendment 3 (August 2018) received the following treatment in each eye:
  Assigned Primary Eye: Selective laser trabeculoplasty (SLT) administered on Day 1 followed by up to three sham bimatoprost SR administrations.
  Contralateral Eye: Sham SLT administered on Day 1 followed by up to three bimatoprost SR 15 µg administrations.
  Bimatoprost SR/sham bimatoprost SR was administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2) and Week 32 (Cycle 3; participants who reached Week 32 prior to implementation of Protocol Amendment 3 only).
- Stage 1: Bimatoprost SR 15 µg (Primary Eye) / SLT (Contralateral Eye): Participants enrolled prior to implementation of Protocol Amendment 3 received the following treatment in each eye:
  Assigned Primary Eye: Sham SLT administered on Day 1 followed by up to three bimatoprost SR 15 µg administrations.
  Contralateral Eye: SLT administered on Day 1 followed by up to three sham bimatoprost SR administrations.
  Bimatoprost SR/sham bimatoprost SR was administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2) and Week 32 (Cycle 3; participants who reached Week 32 prior to implementation of Protocol Amendment 3 only).
- Stage 2: SLT (Primary Eye) / Bimatoprost SR 10 µg (Contralateral Eye): Participants enrolled after implementation of Protocol Amendment 3 received the following treatment in each eye:
  Assigned Primary Eye: SLT administered on Day 1 followed by up to two sham bimatoprost SR administrations.
  Contralateral Eye: Sham SLT administered on Day 1 followed by up to two bimatoprost SR 10 µg administrations.
  Bimatoprost SR/sham bimatoprost SR was administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2). After implementation of Protocol Amendment 6, Cycle 2 retreatment could have occurred after Week 16 and prior to Month 12 based on when retreatment criteria were met.
- Stage 2: Bimatoprost SR 10 µg (Primary Eye) / SLT (Contralateral Eye): Participants enrolled after implementation of Protocol Amendment 3 received the following treatment in each eye:
  Assigned Primary Eye: Sham SLT administered on Day 1 followed by up to two bimatoprost SR 10 µg administrations.
  Contralateral Eye: SLT administered on Day 1 followed by up to two sham bimatoprost SR administrations.
  Bimatoprost SR/sham bimatoprost SR was administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2). After implementation of Protocol Amendment 6, Cycle 2 retreatment could have occurred after Week 16 and prior to Month 12 based on when retreatment criteria were met.
Period: Overall Study
Arm/Group | Stage 1: SLT (Primary Eye) / Bimatoprost SR 15 µg (Contralateral Eye) | Stage 1: Bimatoprost SR 15 µg (Primary Eye) / SLT (Contralateral Eye) | Stage 2: SLT (Primary Eye) / Bimatoprost SR 10 µg (Contralateral Eye) | Stage 2: Bimatoprost SR 10 µg (Primary Eye) / SLT (Contralateral Eye)
Started | 29 | 28 | 92 | 91
Received Treatment (Participants are counted as treated if either eye received study treatment.) | 29 | 27 | 90 | 90
Completed | 24 | 22 | 77 | 78
Not Completed | 5 | 6 | 15 | 13
Not completed — Adverse Event | 3 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 4 | 6 | 6
Not completed — Protocol Violation | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — Screen Failure | 0 | 0 | 1 | 0
Not completed — Other, Not Specified | 0 | 0 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Stage 1: SLT (Primary Eye) / Bimatoprost SR 15 μg (Contralateral Eye): Participants enrolled prior to implementation of Protocol Amendment 3 (August 2018) received the following treatment in each eye:
  Assigned Primary Eye: Selective laser trabeculoplasty (SLT) administered on Day 1 followed by up to three sham bimatoprost SR administrations.
  Contralateral Eye: Sham SLT administered on Day 1 followed by up to three bimatoprost SR 15 μg administrations.
  Bimatoprost SR/sham bimatoprost SR was administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2) and Week 32 (Cycle 3; participants who reached Week 32 prior to implementation of Protocol Amendment 3 only).
- Stage 1: Bimatoprost SR 15 μg (Primary Eye) / SLT Contralateral Eye): Participants enrolled prior to implementation of Protocol Amendment 3 received the following treatment in each eye:
  Assigned Primary Eye: Sham SLT administered on Day 1 followed by up to three bimatoprost SR 15 μg administrations. Contralateral Eye: SLT administered on Day 1 followed by up to three sham bimatoprost SR administrations.
  Bimatoprost SR/sham bimatoprost SR was administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2) and Week 32 (Cycle 3; participants who reached Week 32 prior to implementation of Protocol Amendment 3 only).
- Stage 2: SLT (Primary Eye) / Bimatoprost SR 10 μg (Contralateral Eye): Participants enrolled after implementation of Protocol Amendment 3 received the following treatment in each eye:
  Assigned Primary Eye: SLT administered on Day 1 followed by up to two sham bimatoprost SR administrations.
  Contralateral Eye: Sham SLT administered on Day 1 followed by up to two bimatoprost SR 10 μg administrations. Bimatoprost SR/sham bimatoprost SR was administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2). After implementation of Protocol Amendment 6, Cycle 2 retreatment could have occurred after Week 16 and prior to Month 12 based on when retreatment criteria were met.
- Stage 2: Bimatoprost SR 10 μg (Primary Eye) / SLT (Contralateral Eye): Participants enrolled after implementation of Protocol Amendment 3 received the following treatment in each eye: Assigned Primary Eye: Sham SLT administered on Day 1 followed by up to two bimatoprost SR 10 μg administrations. Contralateral Eye: SLT administered on Day 1 followed by up to two sham bimatoprost SR administrations.
  Bimatoprost SR/sham bimatoprost SR was administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2). After implementation of Protocol Amendment 6, Cycle 2 retreatment could have occurred after Week 16 and prior to Month 12 based on when retreatment criteria were met.
- Total: Total of all reporting groups
Arm/Group | Stage 1: SLT (Primary Eye) / Bimatoprost SR 15 μg (Contralateral Eye) | Stage 1: Bimatoprost SR 15 μg (Primary Eye) / SLT Contralateral Eye) | Stage 2: SLT (Primary Eye) / Bimatoprost SR 10 μg (Contralateral Eye) | Stage 2: Bimatoprost SR 10 μg (Primary Eye) / SLT (Contralateral Eye) | Total
Number analyzed (Participants) | 29 | 28 | 92 | 91 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographic data were analyzed separately for participants in Stage 1 and Stage 2.
  years
    Stage 1: number analyzed (Participants) | 29 | 28 | 0 | 0 | 57
    Stage 1 | 64.9 (12.32) | 59.6 (13.59) |  |  | 62.3 (13.11)
    Stage 2: number analyzed (Participants) | 0 | 0 | 92 | 91 | 183
    Stage 2 |  |  | 62.6 (11.61) | 62.1 (10.74) | 62.4 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 46 | 48 | 122
  Male | 13 | 16 | 46 | 43 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 6 | 10 | 21
  Not Hispanic or Latino | 28 | 24 | 86 | 81 | 219
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 25 | 23 | 58 | 69 | 175
  Black or African American | 1 | 2 | 27 | 14 | 44
  Asian | 3 | 3 | 4 | 6 | 16
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 2
  Not Reported | 0 | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure at Week 4
Description: Intraocular pressure was measured at 8 am (Hour 0) at each visit in each eye using the Goldmann applanation tonometer. A negative change from Baseline indicates a decrease (improvement) in intraocular pressure. A mixed-effects model with repeated measures (MMRM) was used for the analysis. IOP measurements obtained after initiation of non-study IOP-lowering treatment in an eye were excluded from the analysis.
Time Frame: Baseline and Week 4
Population: The intent-to-treat (ITT) population is defined as all randomized participants. Primary efficacy analysis was performed for participants enrolled in Stage 2. Overall Number of Participants / Units Analyzed reflects the number of participants and eyes with data available for the analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Units Other Than Participants: Eyes
Groups:
- Stage 2: SLT: One 360° administration of SLT on Day 1 followed by up to two sham bimatoprost SR administrations.
- Stage 2: Bimatoprost SR 10 µg: Sham SLT on Day 1 followed by bimatoprost SR 10 µg administered on Day 4 with repeat administration at Week 16 or after Week 16 and prior to Month 12 depending on when retreatment criteria were met.
Arm/Group | Stage 2: SLT | Stage 2: Bimatoprost SR 10 µg
Number analyzed (Participants) | 168 | 170
Number analyzed (Eyes) | 168 | 170
mmHg | -6.2 (0.28) | -6.8 (0.28)
Statistical Analysis 1: Comparison: Stage 2: SLT vs Stage 2: Bimatoprost SR 10 µg; Test type: Non-Inferiority — Statistical non-inferiority of Bimatoprost SR 10 µg to SLT was demonstrated if the upper limit of the 95% confidence interval (CI) for the least squares (LS) mean difference between the Bimatoprost SR 10 µg eyes and SLT eyes was ≤ 1.5 mmHg at Weeks 4, 12, and 24. Clinical non-inferiority of Bimatoprost SR 10 µg to SLT was considered if the upper limit of the 95% CI was ≤ 1.0 mmHg at 2 out of the 3 visits of Weeks 4, 12, and 24; p = 0.0231, Mixed Effect Model Repeated Measurement; The model includes treatment, visit, eye, baseline IOP, treatment-by-visit, visit-by-baseline, and visit-by-eyes interactions as covariates; LS Mean Difference = -0.6, 95% CI 2-sided [-1.03 to -0.08], Standard Error of Mean 0.24

2. Primary Outcome: Change From Baseline in Intraocular Pressure at Week 12
Description: Intraocular pressure was measured at 8 am (Hour 0) at each visit in each eye using the Goldmann applanation tonometer. A negative change from Baseline indicates a decrease (improvement) in intraocular pressure. An MMRM was used for the analysis. IOP measurements obtained after initiation of non-study IOP-lowering treatment in an eye were excluded from the analysis.
Time Frame: Baseline and Week 12
Population: The ITT population is defined as all randomized participants. Primary efficacy analysis was performed for participants enrolled in Stage 2. Overall Number of Participants / Units Analyzed reflects the number of participants and eyes with data available for the analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | Stage 2: SLT | Stage 2: Bimatoprost SR 10 µg
Number analyzed (Participants) | 149 | 156
Number analyzed (Eyes) | 149 | 156
mmHg | -6.4 (0.30) | -6.9 (0.30)
Statistical Analysis 1: Comparison: Stage 2: SLT vs Stage 2: Bimatoprost SR 10 µg; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.1615, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.04 to 0.18], Standard Error of Mean 0.31

3. Primary Outcome: Change From Baseline in Intraocular Pressure at Week 24
Description: as for outcome 2
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | Stage 2: SLT | Stage 2: Bimatoprost SR 10 µg
Number analyzed (Participants) | 138 | 145
Number analyzed (Eyes) | 138 | 145
mmHg | -6.5 (0.28) | -6.9 (0.27)
Statistical Analysis 1: Comparison: Stage 2: SLT vs Stage 2: Bimatoprost SR 10 µg; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.1673, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.97 to 0.17], Standard Error of Mean 0.29

4. Secondary Outcome: Time to Initial Use of Non-study IOP-lowering Treatment
Description: The time from the date of initial treatment to the date date of first use of non-study IOP-lowering treatment (rescue) was analyzed using the Kaplan-Meier method.
  If a participant did not use any non-study IOP-lowering treatment in an eye, then the event (initial use of non-study IOP-lowering treatment) time was censored at the study exit date or the last visit date if the study exit date was not available.
Time Frame: From first administration of study treatment to the end of study; overall median follow-up time of 728 days.
Population: Participants in the ITT population enrolled in Stage 2; eyes that received study treatment are included in the analysis.
Measure: Number (95% Confidence Interval); unit: days
Units Other Than Participants: Eyes
Arm/Group | Stage 2: SLT | Stage 2: Bimatoprost SR 10 µg
Number analyzed (Participants) | 180 | 175
Number analyzed (Eyes) | 180 | 175
days
  25% percentile | 263 [167.0 to 329.0] | 276 [217.0 to 323.0]
  50% percentile | NA [736.0 to NA] — Data could not be estimated due to the low number of events. | 732 [496.0 to NA] — Data could not be estimated due to the low number of events.
  75% percentile | NA [NA to NA] — Data could not be estimated due to the low number of events. | NA [NA to NA] — Data could not be estimated due to the low number of events.

5. Secondary Outcome: Percentage of Eyes Achieving ≥ 20% Reduction in IOP From Baseline Regardless of Cycle
Description: Intraocular pressure was measured at 8 am (Hour 0) at each visit in each eye using the Goldmann applanation tonometer.
  For by-cycle analyses, cycle number refers to the administration cycle for bimatoprost SR, or sham bimatoprost SR administration in SLT-treated eyes. For SLT-treated eyes cycle number does not refer to SLT administrations, because SLT was only performed once (Day 1). The Day/Week number refers to the number of days/weeks after bimatoprost SR/sham bimatoprost SR administration.
  IOP measurements obtained after initiation of non-study IOP-lowering treatment in an eye were excluded from the analysis.
Time Frame: Baseline, Day 2, Weeks 4, 8, 12, 15, 20, 24, 28, 31, 36, 40, 44, 47, 52, Months 13, 14, 15, 16, 18, 20, 22, 24
Population: Participants/eyes enrolled in Stage 2 with available IOP data at Baseline and each time point; participants who received retreatment with bimatoprost SR/sham bimatoprost SR at or after Week 16 are not included in Cycle 1 time points from the date of retreatment.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Stage 2: SLT | Stage 2: Bimatoprost SR 10 µg
Number analyzed (Participants) | 183 | 183
Number analyzed (Eyes) | 183 | 183
percentage of eyes
  Day 2: number analyzed (Participants) | 171 | 172
  Day 2: number analyzed (Eyes) | 171 | 172
  Day 2 | 59.1 | 86.6
  Week 4: number analyzed (Participants) | 168 | 170
  Week 4: number analyzed (Eyes) | 168 | 170
  Week 4 | 68.5 | 71.2
  Week 8: number analyzed (Participants) | 164 | 166
  Week 8: number analyzed (Eyes) | 164 | 166
  Week 8 | 64.0 | 75.3
  Week 12: number analyzed (Participants) | 149 | 156
  Week 12: number analyzed (Eyes) | 149 | 156
  Week 12 | 71.1 | 71.8
  Week 15: number analyzed (Participants) | 147 | 152
  Week 15: number analyzed (Eyes) | 147 | 152
  Week 15 | 65.3 | 61.2
  Week 20: number analyzed (Participants) | 145 | 150
  Week 20: number analyzed (Eyes) | 145 | 150
  Week 20 | 62.8 | 67.3
  Week 24: number analyzed (Participants) | 138 | 145
  Week 24: number analyzed (Eyes) | 138 | 145
  Week 24 | 73.2 | 75.2
  Week 28: number analyzed (Participants) | 129 | 133
  Week 28: number analyzed (Eyes) | 129 | 133
  Week 28 | 72.1 | 71.4
  Week 31: number analyzed (Participants) | 126 | 132
  Week 31: number analyzed (Eyes) | 126 | 132
  Week 31 | 67.5 | 62.1
  Week 36: number analyzed (Participants) | 126 | 128
  Week 36: number analyzed (Eyes) | 126 | 128
  Week 36 | 68.3 | 55.5
  Week 40: number analyzed (Participants) | 122 | 121
  Week 40: number analyzed (Eyes) | 122 | 121
  Week 40 | 72.1 | 62.0
  Week 44: number analyzed (Participants) | 116 | 114
  Week 44: number analyzed (Eyes) | 116 | 114
  Week 44 | 65.5 | 57.9
  Week 47: number analyzed (Participants) | 114 | 110
  Week 47: number analyzed (Eyes) | 114 | 110
  Week 47 | 83.3 | 70.9
  Week 52: number analyzed (Participants) | 111 | 110
  Week 52: number analyzed (Eyes) | 111 | 110
  Week 52 | 78.4 | 66.4
  Month 13: number analyzed (Participants) | 78 | 70
  Month 13: number analyzed (Eyes) | 78 | 70
  Month 13 | 73.1 | 65.7
  Month 14: number analyzed (Participants) | 79 | 72
  Month 14: number analyzed (Eyes) | 79 | 72
  Month 14 | 73.4 | 56.9
  Month 15: number analyzed (Participants) | 75 | 67
  Month 15: number analyzed (Eyes) | 75 | 67
  Month 15 | 72.0 | 61.2
  Month 16: number analyzed (Participants) | 82 | 72
  Month 16: number analyzed (Eyes) | 82 | 72
  Month 16 | 76.8 | 70.8
  Month 18: number analyzed (Participants) | 72 | 63
  Month 18: number analyzed (Eyes) | 72 | 63
  Month 18 | 75.0 | 60.3
  Month 20: number analyzed (Participants) | 73 | 61
  Month 20: number analyzed (Eyes) | 73 | 61
  Month 20 | 79.5 | 62.3
  Month 22: number analyzed (Participants) | 70 | 55
  Month 22: number analyzed (Eyes) | 70 | 55
  Month 22 | 78.6 | 69.1
  Month 24: number analyzed (Participants) | 71 | 57
  Month 24: number analyzed (Eyes) | 71 | 57
  Month 24 | 73.2 | 66.7

6. Secondary Outcome: Change From Baseline in IOP at Weeks 8, 15, and 20
Description: IOP was measured at 8 am (Hour 0) at each visit in each eye using the Goldmann applanation tonometer. A negative change from Baseline indicates a decrease (improvement) in intraocular pressure. IOP measurements obtained after initiation of non-study IOP-lowering treatment in an eye were excluded from the analysis.
Time Frame: Baseline and Weeks 8, 15, and 20
Population: Intent-to-treat poulation participants enrolled in Stage 2 with available IOP data at each time point.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | Stage 2: SLT | Stage 2: Bimatoprost SR 10 µg
Number analyzed (Participants) | 183 | 183
Number analyzed (Eyes) | 183 | 183
mmHg
  Baseline | 25.1 (3.00) | 25.2 (2.99)
  Week 8: number analyzed (Participants) | 164 | 166
  Week 8: number analyzed (Eyes) | 164 | 166
  Week 8 | -6.1 (3.52) | -6.8 (3.96)
  Week 15: number analyzed (Participants) | 147 | 152
  Week 15: number analyzed (Eyes) | 147 | 152
  Week 15 | -6.0 (3.58) | -6.0 (4.36)
  Week 20: number analyzed (Participants) | 145 | 150
  Week 20: number analyzed (Eyes) | 145 | 150
  Week 20 | -5.9 (3.44) | -6.4 (3.97)

ADVERSE EVENTS:
Time Frame: All-cause mortality (based on all randomized participants): for an overall median follow-up time of 728 days. Adverse events (AEs; based on all treated participants*): from first dose of study drug up to Month 24 ±7 days. *Six participants who started treatment received SLT only (1 participant had a planned Stage 1 treatment of Bimatoprost SR 15 µg; 5 participants had a planned Stage 2 treatment of Bimatoprost SR 10 µg); these participants are included only in the SLT reporting groups.
Description: Ocular AEs (i.e., those reported for the system organ class 'eye disorders' plus those footnoted as 'ocular events') are reported for the eye that received the treatment specified. Because this is a paired-eye study, and both eyes belong to a single participant, non-ocular AEs affect both reporting groups, and are reported under both interventions.
Groups:
- Stage 1: SLT: Selective laser trabeculoplasty (SLT) administered on Day 1 followed by up to three sham bimatoprost SR administrations.
  Sham bimatoprost SR was administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2) and Week 32 (Cycle 3; participants who reached Week 32 prior to implementation of Protocol Amendment 3 only).
- Stage 1: Bimatoprost SR 15 µg: Sham SLT administered on Day 1 followed by up to three bimatoprost SR 15 µg administrations.
  Bimatoprost SR was administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2) and Week 32 (Cycle 3; participants who reached Week 32 prior to implementation of Protocol Amendment 3 only).
- Stage 2: SLT: SLT administered on Day 1 followed by up to two sham bimatoprost SR administrations.
  Sham bimatoprost SR was administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2; participants who reached Week 32 prior to implementation of Protocol Amendment 3 only).
  Sham bimatoprost SR was administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2). After implementation of Protocol Amendment 6, Cycle 2 retreatment could have occurred after Week 16 and prior to Month 12 based on when retreatment criteria were met.
- Stage 2: Bimatoprost SR 10 µg: Sham SLT administered on Day 1 followed by up to two bimatoprost SR 10 µg administrations.
  Bimatoprost SR was administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2; participants who reached Week 32 prior to implementation of Protocol Amendment 3 only).
  Bimatoprost SR was administered on Day 4 (Cycle 1) and at Week 16 (Cycle 2). After implementation of Protocol Amendment 6, Cycle 2 retreatment could have occurred after Week 16 and prior to Month 12 based on when retreatment criteria were met.
Arm/Group | Stage 1: SLT | Stage 1: Bimatoprost SR 15 µg | Stage 2: SLT | Stage 2: Bimatoprost SR 10 µg
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57 | 2/183 | 2/183
Serious Adverse Events (participants affected / at risk) | 3/56 | 3/55 | 18/180 | 22/175
Other Adverse Events (participants affected / at risk) | 41/56 | 49/55 | 107/180 | 121/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: SLT (N=56) | Stage 1: Bimatoprost SR 15 µg (N=55) | Stage 2: SLT (N=180) | Stage 2: Bimatoprost SR 10 µg (N=175)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CATARACT SUBCAPSULAR (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CORNEAL ENDOTHELIAL CELL LOSS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CORNEAL OEDEMA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CORNEAL THICKENING (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EPISCLERITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RETINAL VEIN OCCLUSION (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BURSITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OESOPHAGEAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PROSTATE CANCER STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
APHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MYELOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VOCAL CORD DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ACCELERATED HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: SLT (N=56) | Stage 1: Bimatoprost SR 15 µg (N=55) | Stage 2: SLT (N=180) | Stage 2: Bimatoprost SR 10 µg (N=175)
ANTERIOR CHAMBER CELL (Eye disorders) | 4 (4) | 6 (8) | 10 (10) | 7 (12)
ANTERIOR CHAMBER FLARE (Eye disorders) | 2 (2) | 4 (4) | 1 (1) | 3 (4)
BLEPHARITIS (Eye disorders) | 3 (3) | 2 (2) | 4 (4) | 3 (3)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 6 (6) | 10 (11) | 2 (2) | 9 (9)
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 13 (22) | 21 (47) | 22 (23) | 35 (48)
CORNEAL ENDOTHELIAL CELL LOSS (Eye disorders) | 4 (4) | 6 (6) | 6 (6) | 11 (13)
CORNEAL TOUCH (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 5 (7) | 7 (10) | 22 (25) | 25 (34)
EYE IRRITATION (Eye disorders) | 4 (4) | 6 (6) | 2 (2) | 4 (4)
EYE PAIN (Eye disorders) | 6 (7) | 6 (11) | 4 (5) | 15 (19)
FOREIGN BODY SENSATION IN EYES (Eye disorders) | 1 (1) | 5 (5) | 2 (2) | 12 (14)
IRITIS (Eye disorders) | 0 (0) | 4 (4) | 0 (0) | 5 (7)
LACRIMATION INCREASED (Eye disorders) | 3 (3) | 1 (1) | 3 (3) | 4 (5)
PHOTOPHOBIA (Eye disorders) | 1 (1) | 5 (8) | 2 (2) | 15 (23)
PUNCTATE KERATITIS (Eye disorders) | 5 (5) | 7 (9) | 19 (25) | 21 (27)
VISION BLURRED (Eye disorders) | 3 (3) | 4 (4) | 4 (4) | 6 (6)
VISUAL FIELD DEFECT (Eye disorders) | 0 (0) | 2 (2) | 18 (22) | 18 (20)
VITREOUS FLOATERS (Eye disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
BRONCHITIS (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 14 (15) | 14 (15)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 9 (10) — ocular event
NASOPHARYNGITIS (Infections and infestations) | 3 (5) | 3 (5) | 8 (8) | 8 (8)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 5 (6) | 8 (8) | 33 (41) | 43 (55) — ocular event
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4) | 2 (2) | 2 (2)
HEADACHE (Nervous system disorders) | 1 (1) | 2 (2) | 10 (10) | 10 (10) — Stage 1 arms = ocular event
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5) | 3 (3) | 3 (3)
HYPERTENSION (Vascular disorders) | 4 (4) | 4 (4) | 15 (16) | 15 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT02507687/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT02507687/SAP_001.pdf